CLINICAL TRIAL: NCT04656860
Title: Encapsulated Fruit and Vegetable Juice Concentrates, Cognition, and Inflammation - A Randomized Placebo-controlled Trial
Brief Title: Juice Plus Supplement Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Alabama, Tuscaloosa (Other)
Collaborators: University of North Texas Health Science Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 17-19-490
Record Dates: First submitted 2020-04-03; First posted 2020-12-07 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2020-06

CONDITIONS: Cognitive Impairment; Alzheimer Disease, Early Onset; Mild Cognitive Impairment
Keywords: Fruits and Vegetables; Inflammation; Cognition
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Inflammation

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to experimental or placebo controlled condition
Who Masked: Participant, Investigator
Masking Description: Both the investigator and the participants will be blinded to study conditions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Juice Plus+ (Experimental): Participants will consume 6 capsules daily consisting of a combination of Juice Plus+ Garden Blend, Juice Plus+ Orchard Blend and Juice Plus+ Berry Blend. Participants will consume supplements for 24-months.
  Interventions: Dietary Supplement: Juice Plus+
- Placebo (Placebo Comparator): Participants will consume 6 capsules daily consisting of microcrystalline cellulose, rice starch, vegetarian capsule (cellulose), and magnesium stearate. Participants in this condition will receive 1-year of supplements after the study is completed.
  Interventions: Dietary Supplement: Juice Plus+

INTERVENTIONS:
Dietary Supplement: Juice Plus+ — Participants will receive encapsulated fruit and vegetable juice concentrates or a placebo for a 24-month period

SUMMARY:
The study is designed to determine whether encapsulated fruit and vegetable juice concentrates can improve biological indicators of cognitive and multiple dimensions of memory and learning.

DETAILED DESCRIPTION:
Preventive interventions that delay the onset of mild cognitive impairment and benign forgetfulness have the potential to delay or even prevent the onset of Alzheimer's disease. However, few studies have examined the feasibility of Encapsulated Fruit and Vegetable Juice Concentrates in robust clinical trials; this limitation prevents investigators from determining the real value of these supplements. Therefore, we propose to enroll 150 adults aged 55 and older to a 24-month randomized placebo-controlled trial. Participants enrolled in the experimental condition will be encouraged to consume 6 Encapsulated Fruit and Vegetable Juice Concentrates capsules per day and 33 grams of a soy-based beverage power per day, which included 5 grams of fiber. Participants enrolled in the controlled condition will receive six placebo capsules and encouraged to maintain an adequate diet. Primary outcomes will include objective measures of cognition, and a panel of inflammatory markers, peptides, enzymes, and other biological markers known to be associated with cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

* • Men and women ≥55 years old will be eligible participants

Exclusion Criteria:

* Prior neurological or psychiatric condition
* Using medications or supplements that influence cognition or inflammation (e.g., nootropics, asprin, and Nonsteroidal anti-inflammatory drugs,),
* Prior cancer diagnosis,
* Major respiratory, kidney, liver, and gastrointestinal issues
* Currently enrolled in a weight loss program or taking an appetite suppressant;
* Current smokers or excessive alcohol users
* Consume >= 4 servings of fruits and vegetables per day

  * Participate in >= 90 minutes of purposeful physical activity per week
  * Do not have a mobile phone
  * Do not have a data plan or regular wireless network

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-03-12 (Actual); Primary Completion 2022-03-12 (Estimated); Study Completion 2023-03-12 (Estimated)

PRIMARY OUTCOMES:
Change in Interleukin -5 | Baseline, Year, 1, and Year 2.
  Interleukin -5 pg/mL
Change in serum Amyloid A | Baseline, Year, 1, and Year 2.
  Serum Amyloid A pg/mL
Change in Interleukin 6 | Baseline, Year, 1, and Year 2.
  Interleukin 6 pg/mL
Change in C-reactive protein | Baseline, Year, 1, and Year 2.
  C-reactive protein pg/mL

SECONDARY OUTCOMES:
Auditory Very Learning Test | Baseline, 6-months, 12-months, 18-months, and 24-months
  Computer automated verbal memory recognition task
Stroop Test | Baseline, 6-months, 12-months, 18-months, and 24-months
  Verbal interference
Trial Making task | Baseline, 6-months, 12-months, 18-months, and 24-months
  Information processing speed

CONTACTS AND LOCATIONS:
Overall Officials: Raheem Paxton, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - University of Alabama, North East Medical Building, Tuscaloosa, Alabama
  - University of Alabama, Tuscaloosa, Alabama

IPD SHARING:
Plan to Share IPD: No
Individual data will not be shared with other researchers